CLINICAL TRIAL: NCT02667639
Title: A Randomized, Double-blind, Placebo-controlled, Single-center, Phase I, Single-dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RPH-104 in Healthy Subjects
Brief Title: Pharmacokinetics and Pharmacodynamics of RPH-104 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: R-Pharm (Industry)
Collaborators: MonitorCRO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RPH104FIH01
Record Dates: First submitted 2016-01-20; First posted 2016-01-29 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2019-09

CONDITIONS: Healthy
Keywords: safety; tolerability; RPH-104; RPH104; Anti-IL1 beta; Anti-IL1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): A single dose of RPH-104 (4, 20, 40, 80 or 160 mg) will be administered subcutaneously.
  Interventions: Biological: RPH-104
- Placebo (Placebo Comparator): A single 0.9% sodium chloride injection will be administered subcutaneously.
  Interventions: Other: Sodium chloride Sterile Injection 0.9% w/v

INTERVENTIONS:
Biological: RPH-104 — Anti-IL-1 Mab
  Arms: Treatment
Other: Sodium chloride Sterile Injection 0.9% w/v — Sterile saline solution
  Arms: Placebo

SUMMARY:
The purpose of this first in human study is to evaluate the safety and tolerability of RPH-104 in humans.

DETAILED DESCRIPTION:
RPH-104 is a macromolecular compound with a molecular weight of 152.715 kilodalton (Data on file) and is capable of binding human interleukin-1 beta (IL-1β). It has also been shown in vitro to be a highly potent inhibitor of IL-1β signalling pathway, with low picomolar inhibitor activity. In this First in Human study, RPH-104 will be evaluated primarily for its safety and tolerability. In a phase I study conducted with health volunteers, a similar monoclonal antibody, canakinumab, was investigated in terms of pharmacokinetics and pharmacodynamics besides efficacy and safety. Similarly, this aimed to investigate effects of RPH-104 on selected pharmacodynamic parameters, including Anti-Drug Antibodies (ADA) along with obtaining first human data on pharmacokinetics of RPH-104 in humans will be investigated in the same study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects.
* Male or female subjects between 18 and 35 years old (inclusive).
* Subject who has normal body weight as determined by a body mass index (BMI) of between 18 kg/m² and 30 kg/m² (inclusive) and within a body weight of ≥50kg and ≤120kg.

Exclusion Criteria:

* Subject who has a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, dermatological, neurological, psychiatric, and hematological or immunological disorder(s), and/or any condition that could constitute a potential safety risk factor or could alter the absorption, distribution, metabolism or elimination of the study drugs.
* Subject who has positive immunoglobulin-M (IgM) antibodies against Epstein-Barr virus (EBV)-viral capsid antigen (VCA) (IgM-anti-EBV-VCA) and Cytomegalovirus (CMV).
* Subject who has a positive Quantiferon TB-Gold (TB) test
* Subject who is positive to Human Immunodeficiency Virus-1/2 antibody (HIV-1/2Ab).
* Subject who has serum hepatitis, or is a carrier of the Hepatitis B surface antigen (HBsAg), or is Hepatitis C virus antibody (HCV-Ab) positive.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2016-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Goksel, MD, PhD, Principal Investigator — ARGEFAR
Locations (1):
- ARGEFAR, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: A single dose of RPH-104 (4, 20, 40, 80 or 160 mg) is administered subcutaneously.
  RPH-104
- Placebo: A single 0.9% sodium chloride injection is administered subcutaneously.
  Sodium chloride Sterile Injection 0.9% w/v
Period: Overall Study
Arm/Group | Treatment | Placebo
Started | 25 | 10
Completed | 25 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects receiving the study medication will be included into the safety evaluation. Subjects who completed the study according to the protocol (per protocol population) will be included into the statistical evaluation. Subject data of drop-out volunteers or volunteers who were not eligible for the study will not be included into statistics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Placebo | Total
Number analyzed (Participants) | 25 | 10 | 35
Age, Customized [Number; unit: participants] — Physical examination, ID check and data entry to study specific Case Report Form.
  participants
    18-35 | 25 | 10 | 10
Sex: Female, Male [Count of Participants; unit: Participants] — Physical examination and data entry to study specific Case Report Form.
  Participants
    Female | 2 | 1 | 3
    Male | 23 | 9 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — Data entry to study specific Case Report Form.
  Participants
    Turkey | 25 | 10 | 35

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Number of participants with study drug related adverse events
Time Frame: Until 60 days after administration
Measure: Number; unit: participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 25 | 10
participants | 0 | 0

2. Primary Outcome: Serious Adverse Events
Description: Number of Participants with Study Drug Related Serious Adverse Events
Time Frame: Until 60 days after administration
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 25 | 10
Participants | 0 | 0

3. Primary Outcome: Respiratory Rate
Description: Percentage of participants with abnormal respiratory rate. The normal respiration rate for an adult at rest is 12 to 20 breaths per minute.
Time Frame: Until 30 days after administration
Measure: Number; unit: percentage of participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 25 | 10
percentage of participants | 0 | 0

4. Primary Outcome: Blood Pressure
Description: Percentage of participants with abnormal blood pressure. An optimal blood pressure level is a reading under 120/80 mmHg
Time Frame: Until 30 days after administration
Measure: Number; unit: percentage of participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 25 | 10
percentage of participants | 0 | 0

5. Primary Outcome: Oxygen Saturation
Description: Percentage of participants with abnormal oxygen saturation. Normal pulse oximeter readings usually range from 95 to 100 percent. Values under 90 percent are considered low.
Time Frame: Until 30 days after administration
Measure: Number; unit: percentage of participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 25 | 10
percentage of participants | 0 | 0

6. Primary Outcome: Body Temperature
Description: Percentage of participants with abnormal body temperature. Among adults, the average body temperature ranges from 97°F (36.1°C) to 99°F (37.2°C).
Time Frame: Until 30 days after administration
Measure: Number; unit: percentage of participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 25 | 10
percentage of participants | 0 | 0

7. Primary Outcome: Clinical Laboratory Tests
Description: Percentage of participants with abnormal clinical laboratory tests. Normal laboratory ranges of the central laboratory were used.
Time Frame: Until 30 days after administration
Measure: Number; unit: percentage of participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 25 | 10
percentage of participants | 0 | 0

8. Secondary Outcome: RPH-104 - Area Under the Curve (AUC)
Description: Mean AUC 0-t (area under the concentration- time curve from time zero to day 30)
Time Frame: Day 1, Day 2, Day3, Day 4, Day 5, Day 6, Day 9, Day 12, Day 15, Day 20, Day 25, Day 30
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 25 | 10
hr*ng/mL
  4 mg | 74500 (24700) | 0 (0)
  20 mg | 430000 (95700) | 0 (0)
  40 mg | 661000 (158000) | 0 (0)
  80 mg | 1610000 (317000) | 0 (0)
  160 mg | 3390000 (1450000) | 0 (0)

9. Secondary Outcome: RPH-104 - Time to Maximum Concentration (Tmax)
Description: Median Tmax. Definition of Tmax is time at which Cmax occurs.
Time Frame: Day 1, Day 2, Day3, Day 4, Day 5, Day 6, Day 9, Day 12, Day 15, Day 20, Day 25, Day 30
Measure: Median (Full Range); unit: hr
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 25 | 10
hr
  4 mg | 96 [94.4 to 192] | 0 [0 to 0]
  20 mg | 96 [48 to 96.2] | 0 [0 to 0]
  40 mg | 120 [96.0 to 192] | 0 [0 to 0]
  80 mg | 96 [72.0 to 120] | 0 [0 to 0]
  160 mg | 120 [72.0 to 120] | 0 [0 to 0]

10. Secondary Outcome: RPH-104 - Elimination Half-life (t1/2)
Description: Mean t½. Definition of t½ is terminal elimination half-life.
Time Frame: Day 1, Day 2, Day3, Day 4, Day 5, Day 6, Day 9, Day 12, Day 15, Day 20, Day 25, Day 30
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 25 | 10
hr
  4 mg | 245 (9.50) | 0 (0)
  20 mg | 249 (6.08) | 0 (0)
  40 mg | 255 (43.1) | 0 (0)
  80 mg | 235 (22.8) | 0 (0)
  160 mg | 243 (40.4) | 0 (0)

11. Secondary Outcome: RPH-104 - Maximum Plasma Concentration (Cmax)
Description: Mean Cmax. Highest concentration determined in the measuring interval.
Time Frame: Day 1, Day 2, Day3, Day 4, Day 5, Day 6, Day 9, Day 12, Day 15, Day 20, Day 25, Day 30
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 25 | 10
ng/mL
  4 mg | 198 (89.1) | 0 (0)
  20 mg | 1280 (402) | 0 (0)
  40 mg | 1650 (257) | 0 (0)
  80 mg | 5120 (1410) | 0 (0)
  160 mg | 10300 (4470) | 0 (0)

ADVERSE EVENTS:
Time Frame: 60 days
Arm/Group | Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/10
Other Adverse Events (participants affected / at risk) | 22/25 | 7/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=25) | Placebo (N=10)
Gastrointestinal disorders (Gastrointestinal disorders) | 8 | 4
Nervous system disorders (Nervous system disorders) | 13 | 4
Infections and infestations (Infections and infestations) | 6 | 3
General disorders and administration site conditions (General disorders) | 3 | 2
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2 | 2
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 | 0
Investigations (Investigations) | 2 | 0
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1 | 1
Cardiac disorders (Cardiac disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Psychiatric disorders (Psychiatric disorders) | 1 | 0
Reproductive system and breast disorders (Reproductive system and breast disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT02667639/Prot_SAP_000.pdf